CLINICAL TRIAL: NCT04931056
Title: Clinical Evaluation of Biomet Microfixation Devices Used in Facial & Mandibular Surgical Procedures. Facial Plating System, HTR PEKK (Midface) and Mandibular Plates: A Post Market Clinical Follow-up Study
Brief Title: A Post Market Clinical Follow-up Study on Biomet Microfixation HTR PEKK (Midface), Facial & Mandibular Plates.
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: 0220-02
Record Dates: First submitted 2021-05-19; First posted 2021-06-18 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Tumor; Facial Fracture; Mandibular Fractures; Fibrous Dysplasia; Osteoma of Mandibular Condyle; Neuroma; Cleft Face; Hemifacial Microsomia; Treacher Collins Syndrome; Miller Syndrome; Nager Syndrome
Keywords: facial plates; mandibular reconstruction; facial reconstruction; condylar tumor; orofacial cleft
MeSH Terms: conditions — Neoplasms; Mandibular Fractures; Fibrous Dysplasia of Bone; Neuroma; Goldenhar Syndrome; Mandibulofacial Dysostosis; Genee-Wiedemann syndrome; Acrofacial dysostosis, Nager type

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Facial Plating: Patients undergoing surgical procedures for facial reconstruction for whom Biomet Microfixation titanium plates (or Ti mini plates) were utilized for the repair.
  Interventions: Device: Titanium Facial Plates
- Mandibular Plating: Patients undergoing surgical procedures for mandibular reconstruction, including TMJ, for whom Biomet Microfixation titanium plates (or Ti mini plates) were utilized for the repair.
  Interventions: Device: Titanium Mandibular Plates; Device: Add-on Condyle
- HTR-PEKK (midface): Patients undergoing surgical procedures for midface reconstruction using custom-made prostheses manufactured on PEEK material.
  Interventions: Device: HTR-PEKK

INTERVENTIONS:
Device: Titanium Facial Plates — The Facial Plating System provides a comprehensive titanium fixation solution for maxillofacial surgery procedures. More than twenty-five different plating options in two systems, the 1.5 mm and 2.0 mm with a variety of instruments, and high torque screws, including meshes, are part of this system. Plates and screws are made of commercially pure titanium per ASTM F-67, Titanium 6Al 4V Alloy per ASTM F-136.
  Other Names: Titanium facial mini plates
  Groups: Facial Plating
Device: Titanium Mandibular Plates — The Mandibular Plating System provides a comprehensive titanium fixation solution for mandibular surgical procedures. Several plating options, a variety of instruments, and high torque screws with various plate shapes are part of this system.
  Plates in the Mandibular Plating System have profiles of various thicknesses. Screws are available in self-tapping, locking and non-locking varieties, and in various sizes between 2.0 mm and 2.3 mm in diameter, and 5 mm to 18 mm in length.
  Other Names: Titanium mandibular mini plates
  Groups: Mandibular Plating
Device: Add-on Condyle — The Add-On Condyle is intended to be implanted in the human jaw to replace the mandibular condyle to functionally reconstruct the temporomandibular joint on a temporary basis for patients undergoing ablative tumor surgery requiring the removal of the native mandibular condyle. This device is not for permanent implantation, traumatic injuries, or for treatment of temporomandibular joint disease.
  Groups: Mandibular Plating
Device: HTR-PEKK — The HTR-PEKK implants are fabricated from polyether-ketone-ketone (PEKK) via selective laser sintering (SLS), a 3D manufacturing technique. The laser sintering machine builds the implant in layers as dictated from a stereolithographic (STL) file of the approved implant. The HTR-PEKK implants are designed individually for each patient to replace bony voids in the facial anatomy using a patient's own CT imaging data. The implant is made to fill an existing or planned void (where appropriate) using computer-aided design technology for anatomy enhancement, correction of trauma injuries, and/or to correct congenital defects in the craniofacial bone.
  Groups: HTR-PEKK (midface)

SUMMARY:
This study will address medical devices manufactured by Biomet Microfixation (d.b.a. Zimmer Biomet) designed for fixation and stabilization of the facial and mandibular skeleton.

DETAILED DESCRIPTION:
The subject devices are:

* plates, screws, and primary instruments from the Biomet Microfixation Facial Plating System, including plates to be specifically used in orthognathic procedures
* plates, screws and primary instruments for the Mandibular Plating System, including and a device intended to temporarily restore the functionality of the temporomandibular joint for patients whose natural condyle has to be resected, subsequent to a tumor ablation ("Add-On Condyle") Additionally, a third device intended for the replacement of bony voids in the facial skeleton will be evaluated in this trial (HTR-PEKK- facial application).

ELIGIBILITY:
Inclusion Criteria:

1. Males or females
2. A patient who underwent one or more of the following surgical procedures completed between January 1, 2015 and December 31, 2019, with plates, screws, and or meshes from the Biomet Microfixation Facial Plating System:

   * Repair of a facial fracture
   * Repair of a facial osteotomy
   * Reconstructive procedures of the facial skeleton
   * Revision procedures where other treatments or devices have failed
3. Available follow-up data at least at 30 days' post-operative

Exclusion Criteria:

1. Active or latent infection at the time of implantation
2. Documented foreign body sensitivity
3. Patients with limited blood supply, insufficient quantity or quality of bone (e.g., osteomalacia or a bone resorption condition such as Paget's disease, osteoporosis, bone metastasis)
4. Patients with documented mental or neurologic conditions who were unwilling or incapable of following postoperative care instructions

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects, who underwent a facial, orbital, or midface procedure and received plates, screws and/or mesh manufactured by Biomet Microfixation. All enrolled subjects will provide data from a retrospective chart review on outcomes of interest.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Survival of implant at 1 year post operative | 1 year
  Frequency and incidence of clinical and radiological adverse events related to the implantation of the subject device leading to removal

SECONDARY OUTCOMES:
Infection rate at 30 days post operative | 30 days
  Implant site infection rate
Allergic reaction related to implant material | up to 2 years
  Clinical and/or pathological assessment of implant allergic reactions leading to removal of the device in the first 2 years post implantation

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sun, PhD, Study Director — Zimmer Biomet
Locations (1):
- San Bernardo Hospital, Salta, Argentina

IPD SHARING:
Plan to Share IPD: No
This data will support regulatory approval on the subject device. Data from this study will not be made available to other researchers